CLINICAL TRIAL: NCT04127747
Title: A Multicenter, Randomized Controlled Clinical Study About Efficacy and Safety of Standard Dose and Individualized Dose of Rituximab in Maintaining Remission in Patients With Moderate to Severe Systemic Lupus Erythematosus
Brief Title: Efficacy of Individualized Rituximab in Maintaining Remission of Moderate and Severe Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-233
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-09

CONDITIONS: Autoimmune Diseases
Keywords: Systemic lupus erythematosus; rituximab
MeSH Terms: conditions — Autoimmune Diseases; Lupus Erythematosus, Systemic | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard dose group (Active Comparator)
  Interventions: Drug: Standard dose of rituximab
- Individualized dose group (Experimental)
  Interventions: Drug: Individualized dose of rituximab

INTERVENTIONS:
Drug: Standard dose of rituximab — Patients in this group will accept RTX 500mg treatment on the first day and on the 6th, 12th,18th and 24th month after that.
  Arms: Standard dose group
Drug: Individualized dose of rituximab — Patients in this group will accept RTX 500mg treatment on the first day of admission. Patients will be followed-up every 3 months, and will receive one RTX 500mg treatment, if CD19 B cell count ≥ 1%, or dsDNA titer increased (dsDNA antibody positive, and increased more than 100% compared with the previous time), or complement C3 level decreased (lower than normal value, and decreased more than 50% compared with the previous time).
  Arms: Individualized dose group

SUMMARY:
Several clinical studies have shown that rituximab is safe and effective for the induction of remission in moderate to severe systemic lupus erythematosus, and has been recommended by several guidelines for the induction of remission in refractory lupus with important organ involvement. However, there are few studies on the use of rituximab in the long-term maintenance and remission of the disease. There is no recognized scheme for the dose, interval and course of treatment of the drug. In this study, patients with moderate and severe systemic lupus erythematosus who achieved remission after standardized treatment were randomly divided into two groups at 1:1 and followed up every 3 months for 24 months. The basic situation and disease activity score of each subject were recorded. The recurrence rate of each observation group was calculated, the influencing factors of disease recurrence were analyzed, and a more reasonable drug use scheme was explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age, 18-65 years old, weight ≥ 40 kg, sex unlimited.
2. Clearly diagnosed with systemic lupus erythematosus.
3. There was at least one BILAG B or above score in the kidney, blood system and nervous system.
4. After standardized treatment with high dose glucocorticoid combined with immunosuppressants such as CTX,MMF or RTX, complete or partial remission of the disease was achieved (up to 1 BILAG B score, and at least 1 BILAG A or BILAG B score less than before).
5. Glucocorticoid: prednisone or the equivalent of prednisone less than or equal to 20 mg daily dose, and can be increased or decreased within 20 mg during the study.
6. Subjects are willing to participate in this study and sign informed consent voluntarily.
7. Prospective subjects agreed to use effective contraception throughout the study period.

Exclusion Criteria:

1. Abnormal liver function: ALT or AST >2ULN，or ALP or TBil >1.5ULN
2. Severe cardiopulmonary disease;
3. Severe blood system disease
4. Patient with malignant tumor;
5. Concurrent infection：Subjects were hospitalized for infection or treated with parenteral antibiotics within 30 days before random; Hepatitis B surface antigen positive or active hepatitis, not treated with hepatitis B antivirus; T-SPOT positive or active tuberculosis, not treated with antituberculous therapy; Any positive in HCV-Ab, HIV-Ab, or TPPA ;
6. Pregnant patients or patients with recent fertility requirements;
7. Received cyclophosphamide treatment within 30 days before random;
8. For any other reason, the investigator believes that it is inappropriate to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease recurrence rate within 24 months. | 24 months
  Evaluate the efficacy of individualized and standard dose rituximab in maintaining remission in moderate to severe SLE patients

SECONDARY OUTCOMES:
Times of use of rituximab in 2 years | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fei Han, Principal Investigator — Zhejiang University; Zhichun Liu, Principal Investigator — The second affiliated hospital of Suzhou University, school of medicine; Wenfeng Tan, Principal Investigator — The people's hospital of Jiangsu province; Xiudi Wu, Principal Investigator — The first hospital of Ningbo; Hongzhi Wang, Principal Investigator — Affiliated Hospital of Jiaxing University; Hongwei Du, Principal Investigator — Jinhua Central Hospital; Yongmei Han, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Second affiliated hospital of zhejiang university，school of medical, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No